CLINICAL TRIAL: NCT02951507
Title: Evaluation of Patient Satisfaction and Biting Force of New Design of Extracoronal Attachment (O T Cap Unilateral Attachment) Versus Conventional Partial Denture for Treatment of Unilateral Mandibular Distal Extension Area
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed mamdouh afify, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: CEBD-CU-2016-10-232
Record Dates: First submitted 2016-10-29; First posted 2016-11-01 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Patient Acceptance of Health Care
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Conventional partial denture (Active Comparator): Intervention will be O T unilateral attachment
  Interventions: Other: O T unilateral attachment
- Conventional removal partial denture (Active Comparator): Intervention will be new design of extra coronal attachment( O T unilateral attachment)
  Interventions: Other: New design of extracoronal attachment system

INTERVENTIONS:
Other: O T unilateral attachment — O T unilateral attachment system
  Arms: Conventional partial denture
Other: New design of extracoronal attachment system — O T unilateral attachment
  Arms: Conventional removal partial denture

SUMMARY:
Comparison of new design of extra coronal castable precision attachment (OT unilateral attachment) and conventional partial denture in patient satisfaction and biting force.

ELIGIBILITY:
Inclusion Criteria:

* patients with unilateral mandibular distal extension area
* Normal crown/root ratio of last premolar
* co-operative patients

Exclusion Criteria:

* completely edentulous patient
* few remaining teeth
* patients exposed to radiotherapy and chemotherapy
* patients with maxillary or mandibular defect

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | 12 months
  OHIP-14 questionnaire

SECONDARY OUTCOMES:
Biting force | 12 months